CLINICAL TRIAL: NCT00661232
Title: An International, Multicenter Trial Assessing Myocardial Viability With Contrast - Enhanced Magnetic Resonance Imaging
Brief Title: Multicenter Myocardial Viability Trial
Status: Completed | Type: Observational
Sponsor: CHI St. Luke's Health, Texas (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Scott D. Flamm, M.D., Principal Investigator, CHI St. Luke's Health, Texas
Other Study IDs: 1102-02-777; NDA# 20-937; IND# 66,506
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Coronary Artery Disease
Keywords: Myocardial Viability; Delayed Enhancement Magnetic Resonance Imaging; Functional Recovery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to test the hypothesis of whether contrast enhanced Magnetic Resonance Imaging can be used to predict improvement of the wall motion in regions of the heart with abnormal movement following bypass surgery or percutaneous angioplasty in various institutions across three continents.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 21 years and < 85 years
* Sinus rhythm
* Weight < 120 kg
* LVEF > 30%
* Wall motion abnormality on Echo. or LV-gram
* Scheduled for revascularization - Angioplasty/Stent or CABG - within 30 days

Exclusion Criteria:

* Resting heart rate > 100 bpm
* Frequent atrial or ventricular ectopy
* Severe aortic stenosis or HOCM
* Unstable angina
* Myocardial infarction within 14 days
* Active congestive heart failure
* Pregnancy
* Known allergy to gadolinium
* Contraindication to MRI

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were recruited from 9 institutions on 3 different continent. All patients recruited for the study had a history of angiographically documented chronic coronary artery disease and resting wall motion abnormalities, and were scheduled for cardiac revascularization (coronary artery bypass surgery or percutaneous intervention).
Sampling Method: Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2003-08-11 (Actual); Primary Completion 2011-01-14 (Actual); Study Completion 2011-05-15 (Actual)

PRIMARY OUTCOMES:
To examine whether the extent of irreversible myocardial injury as assessed by Delayed Enhancement Magnetic Resonance Imaging can predict the extent of functional recovery after revascularization in patients with chronic coronary artery disease (CAD). | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Flamm, M.D., Principal Investigator — CHI St. Luke's Health, Texas
Locations (7):
- United States (2):
  - St. Luke's Episcopal Hospital, Houston, Texas
  - St. Luke's Episcopal Location, Houston, Texas
- Cliniques Universitaires St. Luc, Brussels, Belgium
- Skejby University Hospital, Aarhus N, Denmark
- Hygeia Hospital, Marousi, Greece
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand
- Cardiac MRI Unit, Leeds, United Kingdom